CLINICAL TRIAL: NCT01301365
Title: Autonomic Response During Cystodistension in Patients Suspected of Having Interstitial Cystitis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Assaf-Harofeh Medical Center, Medical Center
Other Study IDs: 178/10
Record Dates: First submitted 2010-12-21; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2010-11

CONDITIONS: Interstitial Cystitis
Keywords: autonomic response
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to check whether patients with cystoscopic findings supporting the diagnosis of Interstitial Cystitis (IC) have a higher autonomic response (change in blood pressure / pulse)than patients without cystoscopic findings.

DETAILED DESCRIPTION:
checking the changes in blood pressure and pulse rate during the initiation of the anesthesia and at the completion of the cystodistension in patient with cystoscopic finding supporting IC

ELIGIBILITY:
Inclusion Criteria:

* All patients having cystodistension suspected of painful bladder syndrome
* symptoms lasting for at least six months
* symptoms suspect of the syndrome: super pubic pain, urinary urgency and frequency
* lack of urinary infection or any other pathology of the urinary tract

Exclusion Criteria:

* Refusal of the patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients having cystodistension suspected of painful bladder syndrome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-04 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
changes in blood pressure and pulse | measuring blood pressure and pulse at the beginning of the anasthesia and at the end of the cystodistension

CONTACTS AND LOCATIONS:
Overall Officials: kobi stav, MD, Study Director — Assaf-Harofeh Medical Center
Locations (1):
- Assaf-HarofehMC, Ẕerifin, Israel